CLINICAL TRIAL: NCT06796075
Title: Identifying Strategies to Reduce Cardiovascular Risk Among Mothers of Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-01959
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Socially Vulnerable Mothers (Experimental): Socially vulnerable mothers of young children, whose children attend formal childcare, will receive telephone-delivered programs over 12 weeks. They will also attend a 6 weeks post-intervention follow-up assessment.
  Interventions: Behavioral: Mom♥Health

INTERVENTIONS:
Behavioral: Mom♥Health — 12-week intervention involving 1) weekly phone calls to mothers regarding education and counseling related to heart healthy lifestyle, as well as strategies for stress reduction; 2) referral to clinical care for identified needs (e.g., elevated blood pressure); and 3) referral to available social resources (e.g., food pantry for identified food insecurity).

SUMMARY:
This single-site research study will pilot-test a context-specific cardiovascular disease (CVD) risk prevention program, Mom♥Health, using two childhood centers at Family Health Centers (FHC) at NYU Langone as platforms for maternal engagement.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a woman
* Is a primary caregiver of child(ren) ≤ 5 years (biological, adopted, fostered) and the child(ren) attends one of the designated childhood centers at FHC at NYU Langone;
* Is between 21-49 years of age
* Is English/Spanish/Mandarin speaking
* Has the capacity and willingness to provide consent

Exclusion Criteria:

* Significant cognitive impairment (evident during screening)
* Current participation in another behavioral clinical trial

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identifies as a woman.
Enrollment: 40 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Complete Intervention Program | Week 12
  Measure of intervention feasibility.
Percentage of Participants who Schedule Clinic/Social Services Appointment for Identified Needs | Week 18
  Measure of intervention feasibility; measured among participants with an identified need.
Client Satisfaction Questionnaire-8 Score | Week 18
  8-item questionnaire related to satisfaction with intervention/service experience. Each item is rated on a Likert scale from 1-4; the total score is the sum of responses and ranges from 8 to 32, with the higher number indicating greater satisfaction.
Percentage of Eligible Mothers who Consent to Enroll | Baseline
  Measure of intervention acceptability.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) Score | Baseline
  The PSS-10 is a 10-item assessment of the degree to which respondents feel that life was overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale. PSS-10 scores range from 0-40, with higher scores indicating greater perceived stress.
Perceived Stress Scale (PSS-10) Score | Week 12
  The PSS-10 is a 10-item assessment of the degree to which respondents feel that life was overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale. PSS-10 scores range from 0-40, with higher scores indicating greater perceived stress.
Perceived Stress Scale (PSS-10) Score | Week 18
  The PSS-10 is a 10-item assessment of the degree to which respondents feel that life was overwhelming, uncontrollable, and unpredictable over the last month. Items are rated on a 5-point scale. PSS-10 scores range from 0-40, with higher scores indicating greater perceived stress.
Patient Health Questionnaire (PHQ-8) Score | Baseline
  The PHQ-8 is an 8-item measure of depressive symptoms during the prior two weeks. Each item has a response scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-24; higher scores indicate greater levels of depression.
Patient Health Questionnaire (PHQ-8) Score | Week 12
  The PHQ-8 is an 8-item measure of depressive symptoms during the prior two weeks. Each item has a response scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-24; higher scores indicate greater levels of depression.
Patient Health Questionnaire (PHQ-8) Score | Week 18
  The PHQ-8 is an 8-item measure of depressive symptoms during the prior two weeks. Each item has a response scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-24; higher scores indicate greater levels of depression.
Mediterranean Eating Pattern for Americans (MEPA) Score | Baseline
  The Mediterranean Eating Pattern for Americans (MEPA) is a 16-item measure of how well a person's diet adheres to the Mediterranean diet. The MEPA score is calculated by assigning a score of 0 or 1 to each item on the MEPA screener. Scores range from 0 to 16; higher scores indicate greater adherence to the Mediterranean diet.
Mediterranean Eating Pattern for Americans (MEPA) Score | Week 12
  The Mediterranean Eating Pattern for Americans (MEPA) is a 16-item measure of how well a person's diet adheres to the Mediterranean diet. The MEPA score is calculated by assigning a score of 0 or 1 to each item on the MEPA screener. Scores range from 0 to 16; higher scores indicate greater adherence to the Mediterranean diet.
Mediterranean Eating Pattern for Americans (MEPA) Score | Week 18
  The Mediterranean Eating Pattern for Americans (MEPA) is a 16-item measure of how well a person's diet adheres to the Mediterranean diet. The MEPA score is calculated by assigning a score of 0 or 1 to each item on the MEPA screener. Scores range from 0 to 16; higher scores indicate greater adherence to the Mediterranean diet.
International Physical Activity Questionnaire (IPAQ) Score | Baseline
  The IPAQ is an assessment how much time participants spent being physically active in the last 7 days. The score is calculated expressed as metabolic equivalent of task (MET)-minutes per week. Higher scores indicate greater physical activity.
International Physical Activity Questionnaire (IPAQ) Score | Week 12
  The IPAQ is an assessment how much time participants spent being physically active in the last 7 days. The score is calculated expressed as metabolic equivalent of task (MET)-minutes per week. Higher scores indicate greater physical activity.
International Physical Activity Questionnaire (IPAQ) Score | Week 18
  The IPAQ is an assessment how much time participants spent being physically active in the last 7 days. The score is calculated expressed as metabolic equivalent of task (MET)-minutes per week. Higher scores indicate greater physical activity.
Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance 8a Score | Baseline
  The PROMIS-Sleep Disturbance subscale is an 8-item questionnaire designed to assess an individual's perception of their sleep disturbances. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 8 to 40, with higher scores indicating more severe sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance 8a Score | Week 12
  The PROMIS-Sleep Disturbance subscale is an 8-item questionnaire designed to assess an individual's perception of their sleep disturbances. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 8 to 40, with higher scores indicating more severe sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance 8a Score | Week 18
  The PROMIS-Sleep Disturbance subscale is an 8-item questionnaire designed to assess an individual's perception of their sleep disturbances. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 8 to 40, with higher scores indicating more severe sleep disturbance.
Mean Blood Pressure | Baseline
  At each time point, 3 BP readings separated by one minute will be obtained. The 3 BP readings will be averaged to obtain the mean study BP.
Mean Blood Pressure | Week 12
  At each time point, 3 BP readings separated by one minute will be obtained. The 3 BP readings will be averaged to obtain the mean study BP.
Mean Blood Pressure | Week 18
  At each time point, 3 BP readings separated by one minute will be obtained. The 3 BP readings will be averaged to obtain the mean study BP.

CONTACTS AND LOCATIONS:
Overall Officials: Milla Arabadjian, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Milla.arabadjian@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Milla.arabadjian@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.